CLINICAL TRIAL: NCT06700369
Title: De-escalation of Neoadjuvant Chemotherapy Regimens (Taxanes Plus Carboplatin Versus Taxanes Only) With Target Therapy Among HER2 Positive Patients
Brief Title: De-escalation of Neoadjuvant Chemotherapy Regimens With Targeted Therapy Among HER2 Positive Patients
Acronym: NacHER2
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z161
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: neoadjuvant chemotherapy; De-escalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Taxanes combined with carboplatin: Taxane (paclitaxel, liposome paclitaxel, docetaxel, albumin paclitaxel), carboplatin combined with trastuzumab and pertuzumab, 6 cycles in total
- Taxanes: Taxane (paclitaxel, liposome paclitaxel, docetaxel, albumin paclitaxel) with trastuzumab and pertuzumab, 6 cycles in total

SUMMARY:
Neoadjuvant therapy is currently the standard treatment process for locally advanced breast cancer, especially for human epidermal growth factor receptor 2 (HER2) positive and triple negative breast cancer, which meets the requirements of tumor ≥ 2cm and/or lymph node positive, and the guidelines recommend neoadjuvant therapy as the first choice. Chemotherapy combined with trastuzumab and pertuzumab is the standard neoadjuvant therapy for HER2 positive breast cancer patients. Taxane plus carboplatin (TCb) is the first choice of chemotherapy recommended by major guidelines; As an alternative, single drug Taxane (T) is also listed as class I recommendation in the latest CSCO guidelines, but the level of evidence is slightly insufficient. Considering the defects such as large side effects of combined chemotherapy, whether single drug chemotherapy can be used as the first choice for some people under the support of targeted drugs remains to be studied.

This project plans to a cohort study, based on the large sample breast disease cohort database established by the breast center of Peking University People's Hospital, and retrospectively include the patients with clinical stage T2 and above and/or lymph node positive breast cancer who received neoadjuvant therapy (TCbHP or THP) from January 1, 2015 to December 31, 2024. Patients of the same type were prospectively included from January 1, 2025 to December 31, 2028. The effectiveness and safety of TCbHP and THP as a neoadjuvant therapy were compared.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with HER2 positive breast cancer diagnosed by biopsy in Peking University People's Hospital;
* 2) The clinical stage was stage II or stage III (i.e. T2 and above, and/or lymph node positive, without distant organ metastasis);
* 3) Received treatment in our hospital and had hospitalization records;
* 4) Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

* 1) Lack of clinical and pathological data (such as imaging data and pathological data);
* 2) Patients with metastatic breast cancer or bilateral breast cancer;
* 3) At the same time, they received anti-tumor therapy in other clinical trials, including endocrine therapy and targeted therapy;
* 4) Receiving other regimens besides the established neoadjuvant regimens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HER2 positive breast cancer patients who received neoadjuvant chemotherapy based on taxanes with trastuzumab, pertuzumab target therapy
Sampling Method: Probability Sample
Enrollment: 519 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
pathology complete response | 6 months
  Postoperative pathology confirmed that the primary breast lesions and axillary lymph nodes had no residual invasive tumor cells (ypT0/is and ypN0)

SECONDARY OUTCOMES:
Invasive disease free survival | 5 years
  the time from study enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.
Disease free survival | 5 years
  the time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.
Breast cancer specific survival | 5 years
  time from study enrollment to death due to breast cancer.
Overall survival | 5 years
  the time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China